CLINICAL TRIAL: NCT06128707
Title: Vestibulo-Ocular Reflex Function in Individuals With Chronic Motion Sensitivity Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 5230167
Record Dates: First submitted 2023-10-25; First posted 2023-11-13 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Motion Sickness
Keywords: Chronic motion sensitivity
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Motion sensitivity group: Participants with a self-reported history of chronic motion sensitivity and who scored greater than or equal to the 30th percentile on the Motion sickness susceptibility questionnaire short form.
- Non-Chronic Motion sensitivity Group: Participants without a self-reported history of chronic motion sensitivity and who scored less than or equal to the 25th percentile on the Motion sickness susceptibility questionnaire short form.

SUMMARY:
Chronic motion sensitivity refers to a sensation of unwellness caused by physical or discerned motion and has a prevalence of 28% in the general population and it is more common in women (27.3%) compared to men.

The investigators theorize that individuals with chronic motion sensitivity will have an impaired inner ear reflex and will be less physically active. Hence, the purpose of this study is to;

1. Determine whether the function of an inner ear reflex is different between young adults with/without chronic motion sensitivity
2. Assess relationships between reflex function and balance in young adults with/without CMS
3. Assess relationships between physical activity and balance in young adults with/without CMS.

DETAILED DESCRIPTION:
Chronic motion sensitivity (CMS), also known as motion sickness, refers to a sensation of unwellness caused by physical or discerned motion. CMS has a prevalence of 28% in the general population and it is more common in women (27.3%) compared to men.

Based on established evidence that individuals with chronic motion sensitivity demonstrate impaired postural stability with vestibular system impairment adjudged to be an inciting stimulus for chronic motion sensitivity, and individuals who practiced more physical and sporting activities have less motion sickness susceptibility than individuals who did not, the investigators theorize that individuals with chronic motion sensitivity will have an impaired inner ear reflex, causing them to be more reliant on other sensory systems like their muscles and joints, and their vision, we also theorize that individuals who are physically active will be less susceptible to chronic motion sensitivity.

The purpose of this study is to;

1. Determine whether the function of an inner ear reflex is different between young adults with/without chronic motion sensitivity
2. Assess relationships between reflex function and balance in young adults with/without CMS
3. Assess relationships between physical activity and balance in young adults with/without CMS.

Participants between the age of 20 and 40 with and without a self-reported history of chronic motion sensitivity (i.e, experiencing nauseousness and/or dizziness during while using various means of transportation such as, car, train, bus, boat, and airplane and/or, recreational fun-fair rides and/or when exposed to conflicting visual images). Participants will be excluded if they report a medical diagnosis of central nervous system disorder, impaired cervical spine range of motion, migraines, seizure disorder, vestibular dysfunction, or any musculoskeletal dysfunction that can limit their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40
* With and without a history of CMS

Exclusion Criteria:

* CNS disorder
* Impaired cervical spine ROM
* Migraines
* Seizures
* Vestibular dysfunction
* Musculoskeletal dysfunction
* Medications causing dizziness

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Participants will be recruited from Loma Linda University and surrounding communities. The study will be conducted in the Loma Linda University Physical Therapy Department's Neuroscience Research Laboratory. Participants between the age of 20 and 30 with and without a self-reported history of chronic motion sensitivity (i.e, experiencing nauseousness and/or dizziness during while using various means of transportation such as, car, train, bus, boat, and airplane and/or, recreational fun-fair rides and/or when exposed to conflicting visual images)
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Bertec vision advantage | 1 day
  Scores on 4 parametters- Baseline visual acuity (Logarithm of the minimum angle of resolution LogMAR)- A measure of optotype size with lower values signifying smaller optotype size and better vision with the head static, Visual processing time (Mili seconds) this is the time taken to identify the size of the optotype, Dynamic visual acuity (Logarithm of the minimum angle of resolution LogMAR)-A measure of optotype size with lower values signifying smaller optotype size and better vision with the head dynamic, Gaze stability test (Degrees per second), this is the highest speed at which the participant can identify the optotype while the head is moving.
Computerized dynamic posturography with immersion virtual reality | 1 day
  Average scores under 2 conditions- Condition one- Eye open, Stable platform, Condition 2 Eye open, sway referenced platform. Each condition measured gives a score known as the equillibrum score measured as age matched normative data with higher scores signifying stronger balance , and a lower scores signifying weaker balance

SECONDARY OUTCOMES:
International Physical activity questionaire short form | 1 day
  Questionaire to assess physical activity

OTHER OUTCOMES:
Motion sickness susceptibility questionnaire short form | 1 day
  Questionnaire used to asses motion sickness susceptibility

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided